CLINICAL TRIAL: NCT03244176
Title: Feasibility Study of Induction and Maintenance Avelumab Plus R-CHOP in Patients With Diffuse Large B Cell Lymphoma (DLBCL): The AvR-CHOP Study
Brief Title: Feasibility Study of Induction and Maintenance Avelumab Plus R-CHOP in Patients With Diffuse DLBCL: The AvR-CHOP Study
Acronym: AvR-CHOP
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Austin Health (Other Government)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Dr. Eliza Hawkes, Chief Principal Investigator, Austin Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS100070-0068
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Lymphomas Non-Hodgkin's B-Cell
Keywords: DLBCL
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label (Other): Avelumab - Single-arm open label study
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — All participants will receive the following treatment:
  Induction phase Avelumab at a dose of 10 mg/kg as a 1hour intravenous (IV) infusion once every 2 weeks for 2 cycles Plus Rituximab at a dose of 375mg/m2 as an IV infusion over at least 1 hour once every 2 weeks for 2 treatments
  Then:
  RCHOP - All participants will receive RCHOP chemotherapy treatment for 6 cycles. Each cycle will last for 21 days. Rituximab, cyclophosphamide, doxorubicin, and vincristine are given on the first day of each cycle by intravenous infusion. Prednisone is given orally from Day 1 until Day 5 of each cycle.
  Then:
  Maintenance phase - All participants will receive Avelumab at a dose of 10 mg/kg as a 1hour intravenous (IV) infusion once every 2 weeks for 6 cycles.
  Other Names: MSB0010718C

SUMMARY:
To evaluate the feasibility of adding induction and maintenance Avelumab to the standard combination of R-CHOP in patients with stage II, III and IV diffuse large B cell lymphoma (DLBCL)

DETAILED DESCRIPTION:
The rationale and primary objective is to evaluate the feasibility of adding induction and maintenance Avelumab into the standard Rituximab, Cyclophosphamide, Doxyrubicin, Vincristine and Prednisolone (RCHOP) regimen in order to examine the effect of programmed death-ligand 1(PDL1) inhibition in patients with stage II, III and IV DLBCL.

Primary endpoint:

• Immune related toxicity which requires discontinuation of Avelumab.

Secondary endpoints:

* Response rates (according to the Lugano classification for Response Criteria for NonHodgkin Lymphoma);
* Failure free survival;
* Overall survival;
* Overall toxicity of treatment (according to CTCAE v 4.0).

Methodology:

All patients (n=28) will receive Avelumab and rituximab 2 weekly for 2 cycles, then RCHOP chemotherapy 3 weekly for 6 cycles then Avelumab 2 weekly for 6 cycles.

The sequential treatment schedule has been designed for several reasons: concurrent Avelumab and RCHOP might result in reduced efficacy of Avelumab owing to the high dose prednisolone component of RCHOP; immune related toxicities of Avelumab given concurrently with RCHOP might result in chemotherapy dose delays and reduced chemotherapy efficacy; the Avelumab plus rituximab prephase will allow for the preliminary assessment of nonchemotherapy agents Avelumab plus rituximab in treatment naïve patients.

Assessments:

* Patients will be reviewed at baseline and prior to each cycle of treatment for toxicity
* Positron emission tomography-computed tomography (PET/CT) will be performed at baseline, after induction phase, after cycle 2 RCHOP, at end of Avelumab (Av) RCHOP and at end of maintenance phase Avelumab.
* Following completion of treatment, patients will be followed up for a total of 5 years (at 3,6,9,12,18,24,36,48 and 60 months posttreatment). No formal routine imaging will be performed during follow up. In patients with relapse, follow up only for survival will be every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects aged 18 years.
2. Histologically proven CD20-positive diffuse large B cell non-Hodgkin lymphoma (DLBCL) according to the current World Health Organization classification including all morphological variants.
3. No previous treatment for lymphoma including chemotherapy, radiotherapy or other investigational drug.
4. Stage II, III and IV disease (Ann Arbor criteria) (must be able to undergo PET/CT imaging for staging purposes.)
5. Eastern Collaborative Oncology Group performance status 0, or 1, unless attributable to lymphoma in which case patients of performance status 2 are also eligible.
6. Adequate bone marrow function with platelets > 100x109/l; neutrophils > 1.5x109/l at the time of study entry unless attributed to bone marrow infiltration by lymphoma.
7. Adequate renal function defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
8. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 × upper limit of institutional normal range unless attributed to lymphoma.
9. Patients must have an acceptable left ventricular ejection fraction (LVEF) i.e. within the local normal range for multigated acquisition scan (MUGA) or ≥ 45% on echocardiogram
10. No concurrent uncontrolled medical condition as determined by the investigator.
11. Life expectancy > 3 months.
12. Negative blood pregnancy test at screening for women of childbearing potential. Effective contraception for both male and female subjects if the risk of conception exists.
13. Signed written informed consent before any trial-related procedure is undertaken that is not part of the standard patient management.

Exclusion Criteria:

1. T-cell lymphoma, transformed follicular lymphoma, grade 3B Follicular lymphoma.
2. Previous history of treated or non-treated indolent lymphoma. However, patients not previously diagnosed with an indolent lymphoma, who have diffuse large B-cell lymphoma with some small cell infiltration in bone marrow or lymph node may be included after consultation with the sponsor.
3. Central nervous system, meningeal or spinal cord involvement by lymphoma.
4. Prior therapy with any antibody or drug targeting T-cell coregulatory proteins (immune checkpoints) such as PD-1, PD-L1, or cytotoxic T-lymphocyte antigen-4 (CTLA-4).
5. Patients with active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

i) Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible ii) Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day iii) Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable.

f) Subjects with a condition requiring systemic treatment with either corticosteroids (> 15 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 15 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

g) Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI-CTCAE v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma) h) Past history of interstitial lung disease. i) Prior organ transplantation, including allogeneic stem-cell transplantation j) Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

k) Neurological contra-indication to vincristine (e.g. pre-existing diabetic neuropathy >grade 1) l) Major surgery for any reason, except diagnostic biopsy, within 4 weeks of enrolment and/or if the subject has not fully recovered from the surgery within 4 weeks of enrolment m) Any other serious active disease, including but not limited to; i) pregnancy or lactation, ii) clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina pectoris, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious cardiac arrhythmia requiring medication (including QTc prolongation of > 470 ms and/or pacemaker) or prior diagnosis of congenital long QT syndrome.

iii) or, uncontrolled active infection, iv) or, uncontrolled diabetes (e.g., hemoglobin A1c ≥ 8%) n) Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS), Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive) o) Medical or psychiatric conditions that compromise the patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Immune-related toxicity | 12 months
  Immune-related toxicity which requires discontinuation of Avelumab

SECONDARY OUTCOMES:
Response Rate | 2 years
  Response Rate to Avelumab + RCHOP according to the Lugano classification for Response Criteria for Non-Hodgkin Lymphoma
Failure Free Survival | 2 years
  Duration of survival without additional systemic therapy, relapse or non-relapse mortality
Overall Survival | 2 years
  Duration of patient survival
Overall Toxicity of Treatment | 12 months
  Overall toxicity as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Hawkes, MD, Principal Investigator — Austin Health
Locations (3):
- Australia (3):
  - Ballarat Health, Ballarat, Victoria
  - Eastern Health, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: Undecided
IPD is the property of the Sponsor (Austin Health). Results from the research intends to be published/presented in relevant publications/conferences for colleague review